CLINICAL TRIAL: NCT02639520
Title: A Double-blind, Controlled, Parallel-group, Randomized, Multicenter Clinical Trial to Assess the Efficacy and Safety of a Herbal Drug Containing Centaury, Lovage Root and Rosemary Leaf (CLR) in Comparison to Fosfomycin Trometamol for the Treatment of Acute Lower Uncomplicated Urinary Tract Infections (uUTIs) in Women
Brief Title: Efficacy of CLR Compared to Fosfomycin Trometamol in Acute Lower uUTIs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bionorica SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CanUTI-7
Record Dates: First submitted 2015-12-11; First posted 2015-12-24 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Urinary Tract Infection
Keywords: Uncomplicated urinary tract infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Fosfomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Canephron® N (Active Comparator): Canephron® N & fosfomycin trometamol-placebo
  Interventions: Drug: Canephron® N; Drug: Fosfomycin trometamol-placebo
- Group Fosfomycin Trometamol (Active Comparator): Canephron® N-placebo & fosfomycin trometamol
  Interventions: Drug: Fosfomycin trometamol; Drug: Canephron® N-placebo

INTERVENTIONS:
Drug: Canephron® N — 2 tablets 3 times a day for 7 days
  Arms: Group Canephron® N
Drug: Fosfomycin trometamol — 1 sachet of 8 g of granules; one single dose on Day 1
  Arms: Group Fosfomycin Trometamol
Drug: Canephron® N-placebo — 2 tablets 3 times a day for 7 days
  Arms: Group Fosfomycin Trometamol
Drug: Fosfomycin trometamol-placebo — 1 sachet of 8 g of granules; one single dose on Day 1
  Arms: Group Canephron® N

SUMMARY:
To demonstrate non-inferiority of a non-antibiotic therapy with CLR versus an antibiotic treatment with fosfomycin trometamol in women suffering from acute lower uUTIs as measured by the proportion of patients who received an additional antibiotic treatment for acute lower uUTIs during the trial.

DETAILED DESCRIPTION:
The trial is designed as a comparison of two different modes of action in order to look for alternatives to antibiotic treatment of uncomplicated UTIs. Treatment with CLR is a nonantibiotic therapy and is compared to an antibiotic treatment. Thus, the trial aim is to reduce antibiotics use and moreover to reduce the pressure of developing bacterial resistance against antibiotics due to widespread use, which is an additional advantage of the CLR therapy.

The trial results are expected to demonstrate that antibiotic prescriptions in women for treatment of lower uUTIs can be reduced by an alternative and safe non-antibiotic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent (IC) and data protection declaration
2. Female outpatients aged 18 to 70 years
3. Sum-score of the main uUTI symptoms (dysuria, pollakisuria, and urgency) reported on the Acute Cystitis Symptom Score (ACSS)-"Typical" domain at Visit 1 is ≥6
4. Symptoms of the acute episode of lower uUTI are developed within not more than 6 days prior to Visit 1
5. Leukocyturia at Visit 1, confirmed by positive dipstick
6. Patients willing to refrain from consuming prohibited concomitant medications and products
7. Non-lactating female patients who are surgically sterile (have had a documented sterilization, bilateral oophorectomy at least 3 months before the start of the trial and/or hysterectomy), or postmenopausal (cessation of menses for at least 12 months), or women of childbearing potential with a negative pregnancy test at Visit 1 willing to use highly effective (failure rate less than 1% per year, i.e., Pearl Index <1) contraception methods, e.g., contraceptive patch, oral, injected or implanted hormonal methods of contraception, during the trial including the follow-up period.

Exclusion Criteria:

1. Any signs of complicated urinary tract infections (UTIs), pyelonephritis (i.e., fever T ≥38.0°C [grade 2], flank and/or back pain, chills and shivers), and/or vulvo-vaginitis with vaginal and/or with urethral discharge (without urination) at Visit 1.
2. Any conditions that may lead to complicated infections (i.e., renal diseases, urinary tract abnormalities or past urinary surgery, urine catheterization, uncontrolled diabetes mellitus, spinal cord injury, etc.).
3. Chronic infection of the urinary tract known from medical history.
4. Persisting signs or symptoms of severe, progressive, or uncontrolled systemic disease (i.e., renal, hepatic, biliary, hematological, gastro-intestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease).
5. Uncontrolled hypertension (a diastolic blood pressure >95 mmHg at Visit 1).
6. Known severe cardiac insufficiency, coronary heart disease, valvular heart disease, cardiac arrhythmia, QT interval prolongation or other severe cardiac disease at Visit 1.
7. Any antibiotic therapy within 30 days prior to Visit 1.
8. Other acute infections (except uUTIs) requiring antibiotic treatment at Visit 1.
9. Patients receiving treatment for suspected or confirmed UTI (antibiotic or phytopharmaceutical) within 30 days prior to Visit 1.
10. Patients who took anti-inflammatory drugs (e.g., ibuprofen) or spasmolytics for any reason within 24 hours prior to Visit 1, and/or are not willing to stop the intake of any of the medication not permitted for use during the trial.
11. Known severe impaired renal function (creatinine clearance <20 mL/min).
12. Active peptic ulcers.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 659 (Actual)
Dates: Start 2015-12; Primary Completion 2017-06 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Intake of any additional antibiotic medication for acute lower uUTIs between Visit 1 and Visit 4 | within 38 days after Visit 1 (=day 1)
  For patients with consistent or worsening of acute lower uUTI symptoms during the trial the investigator may offer an additional antibiotic therapy at any post-baseline visit. In this case, the patient will be considered a "treatment failure" due to lack of efficacy of the IMP. The alternative antibiotic therapy offered to the patient and the reason for the alternative therapy (i.e., persisting or recurrent symptoms) is to be documented.
  The primary variable for the assessment of efficacy is the proportion of patients who received additional antibiotic treatment for acute lower uUTI between Visit 1 and Visit 4 (defined as AB-rate).

CONTACTS AND LOCATIONS:
Overall Officials: Florian Wagenlehner, Prof., Principal Investigator — Universitätsklinikum Gießen und Marburg GmbH
Locations (1):
- Justus-Liebig-Universität, Giessen, Hesse, Germany

REFERENCES:
- [Derived] Wagenlehner FM, Abramov-Sommariva D, Holler M, Steindl H, Naber KG. Non-Antibiotic Herbal Therapy (BNO 1045) versus Antibiotic Therapy (Fosfomycin Trometamol) for the Treatment of Acute Lower Uncomplicated Urinary Tract Infections in Women: A Double-Blind, Parallel-Group, Randomized, Multicentre, Non-Inferiority Phase III Trial. Urol Int. 2018;101(3):327-336. doi: 10.1159/000493368. Epub 2018 Sep 19. PMID 30231252